CLINICAL TRIAL: NCT04017260
Title: Combined Open and Closed Approach for Management of Pilonidal Sinus by Special U-shaped Sutures Without Drain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, clinical professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zagazig university
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal sinus, combined, sutures, drain
MeSH Terms: conditions — Pilonidal Sinus | interventions — Open Abdomen Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- open and closed technique (Experimental): treatment of pilonidal sinus by open and closed approach
  Interventions: Procedure: open and closed approach
- Rhomboid flap technique (Experimental): treatment of pilonidal sinus by Rhomboid flap
  Interventions: Procedure: Rhomboid flap technique
- karydakis technique (Experimental): treatment of pilonidal sinus by Karydakis
  Interventions: Procedure: Karydakis technique
- open technique (Experimental): treatment of pilonidal sinus by open approach
  Interventions: Procedure: open technique

INTERVENTIONS:
Procedure: open and closed approach — The patients were hospitalized, and the site of the operation was shaved on the day of the surgery. All Patients were operated on under spinal anesthesia. Antibiotic was administered to all patients as prophylaxis 60 minutes prior to the surgery. An adhesive tape was used to part the buttocks. The patients were placed in the jack-knife position. (Fig. 1). Methylene blue was injected without pressure through the external opening to delineate the sinus. The operation site was cleaned with 10% povidone-iodine. All sinus tracts were resected en bloc via elliptical incision down to presacral fascia with meticulous hemostasis.
  Group A:The wound was closed with 0 polypropylene u-shaped sutures .
  Arms: open and closed technique
Procedure: Rhomboid flap technique — The patients were hospitalized, and the site of the operation was shaved on the day of the surgery. All Patients were operated on under spinal anesthesia. Antibiotic was administered to all patients as prophylaxis 60 minutes prior to the surgery. An adhesive tape was used to part the buttocks. The patients were placed in the jack-knife position. (Fig. 1). Methylene blue was injected without pressure through the external opening to delineate the sinus. The operation site was cleaned with 10% povidone-iodine. All sinus tracts were resected en bloc via elliptical incision down to presacral fascia with meticulous hemostasis.Rhomboid flap technique: involve closure of the defect after excision of all sinuses with Rhomboid flap of skin and subcutaneous tissue
  Arms: Rhomboid flap technique
Procedure: Karydakis technique — The patients were hospitalized, and the site of the operation was shaved on the day of the surgery. All Patients were operated on under spinal anesthesia. Antibiotic was administered to all patients as prophylaxis 60 minutes prior to the surgery. An adhesive tape was used to part the buttocks. The patients were placed in the jack-knife position. (Fig. 1). Methylene blue was injected without pressure through the external opening to delineate the sinus. The operation site was cleaned with 10% povidone-iodine. All sinus tracts were resected en bloc via elliptical incision down to presacral fascia with meticulous hemostasis.the long axis of the ellipse is parallel to the midline and 2cm from it.undercutting incision is made along the whole length 1cm below the skin surface then unrolling the flap over the midline.
  Arms: karydakis technique
Procedure: open technique — The patients were hospitalized, and the site of the operation was shaved on the day of the surgery. All Patients were operated on under spinal anesthesia. Antibiotic was administered to all patients as prophylaxis 60 minutes prior to the surgery. An adhesive tape was used to part the buttocks. The patients were placed in the jack-knife position. (Fig. 1). Methylene blue was injected without pressure through the external opening to delineate the sinus. The operation site was cleaned with 10% povidone-iodine. All sinus tracts were resected en bloc via elliptical incision down to presacral fascia with meticulous hemostasis.Open procedure involved a wide excision of the pilonidal sinus tract and healing by secondary intention.
  Arms: open technique

SUMMARY:
Introduction: Pilonidal sinus disease (PSD) is a common surgical disease frequently seen in the intergluteal cleft. The treatment of this problem is mainly surgical.

Aim: introduce a novel technique of combined open and closed approach for management of primary pilonidal sinus (non-recurrent) by special U-shaped sutures and compare it with other techniques as regard operative time, time of complete wound healing, postoperative pain , time to stop analgesic drugs and evaluate the result of surgery without drain.

Patients: this study was conducted on 160 patients with PSD in the sacrococcygeal region who underwent operation between December 2015 and December 2017. All cases are divided randomly into four groups each consists of 40 patients.

DETAILED DESCRIPTION:
1. Introduction Pilonidal sinus disease (PSD) is a common disease seen in the intergluteal cleft. This disease is usually seen between the ages of 15 years and 35 years, and males are affected more often than females [1]. The incidence of the disease is 26/100,000 in the general population [2]. The most accepted theory for this disease development is the penetration of shed hair into the skin and is associated with inflammation, abscess and sinus formation [1]. The depth of the intergluteal sulcus, the number of loose hair, and the stiffness of the hairs play important role in the disease etiology [3]. The reason for the wide acceptance of the acquired theory may be the high recurrence rates of up to 30% even after the most radical local excisions of pilonidal disease, which suggests that a pilonidal sinus is an acquired new disease rather than the persistence of some existing sinuses [4]. Although many medical and surgical methods have been proposed for this disease management, no clear consensus about the best method of treatment has been reported so far in the literature. Medical treatment modalities include phenol, silver nitrate, and electro cauterization of the cavity .The surgical options include excising the sinus to the level of the sacrococcygeal fascia and primary closure, or leaving it to secondary healing, Z-plasty, split-skin grafting, Rhomboid flap rotation, or Karydakis flap [5]. Eradication of the pilonidal sinus through wide surgical excision is still the cornerstone of treatment, yielding good long-term results, but at the expense of postoperative complications, prolonged hospital stay and a period of off-work up to 4-8 weeks, substantial pain, sub-optimal aesthetic results and recurrence [6].

   The main problem after PSD surgery is recurrence, and recurrence rates have been reported in the literature to range from 3% to 46%, depending on the technique used [7].

   The aim of the present study was to analyze , evaluate and compare the short term and long term clinical results of this novel technique of combined closed and open approach for management of pilonidal sinus by special U-shaped sutures without drain, Rhomboid flap technique, Karydakis technique and open technique, an approach that allows surgeons to overcome these techniques complications.
2. Materials and methods This is a controlled clinical trial on 160 patients who had been operated on for PSD between December 2015 and December 2017 in faculty of medicine, Zagazig University, after approval from medical ethical committee. Fifteen patients were lost during the study as we cannot reach them by any way and were excluded from the study. The remaining consecutive patients were included in this prospective analysis.

   The patients were divided into 4 groups: Group A: 40 patients underwent combined open and closed technique, Group B: 40 patients underwent Rhomboid flap technique, Group C: 40 patients underwent Karydakis technique and Group D: 40 patients underwent open technique and wound is left to heal with secondary intention. Patients are grouped randomizally that patient 1 went to group A and patient 2 went to group B and patient 3 went to group c and patient 4 went to group D and the process is repeated.

   Time of operation, postoperative morbidity and hospital stay, and loss of work days, duration of wound healing and recurrence were analyzed. Informed consent was obtained from all individual participants included in the study.

   Inclusion criteria include primary PSD in intergluteal region between 18-35 years. Also those fulfilling the diagnostic criteria of Chronic discharging sinus/sinuses in natal cleft with or without surrounding tissue inflammation and with associated pain and bleeding on clinical evaluation were also included in our study. Exclusion criteria include recurrent pilonidal sinus, patients who were terminally ill, had Uncontrolled diabetics, were Immunocompromised and immunosuppressed patients, had acute pilonidal abscess.

   The patients with PSD underwent the procedure by the same surgeon. Infected sinuses were treated with antibiotics prior to the surgery for at least 2 weeks.

   The patient's age, sex, operation time, mean hospital stay, postoperative wound complications, cosmetic appearance and recurrence rate, and hypoesthesia in the gluteal region were recorded during follow-up period. Clinical assessments were performed postoperatively on the 1st day, 3rd day, 7th day, and 10th day and by telephone on the 1st month, 3rd month, 6th month, and 12th month.

   2.1. Operative technique The patients were hospitalized, and the site of the operation was shaved on the day of the surgery. All Patients were operated on under spinal anesthesia. Antibiotic was administered to all patients as prophylaxis 60 minutes prior to the surgery. An adhesive tape was used to part the buttocks. The patients were placed in the jack-knife position. (Fig. 1). Methylene blue was injected without pressure through the external opening to delineate the sinus. The operation site was cleaned with 10% povidone-iodine. All sinus tracts were resected en bloc via elliptical incision down to presacral fascia with meticulous hemostasis. (Fig 2)(Fig.3).

   Group A:The wound was closed with 0 polypropylene sutures including skin, subcutaneous tissue and including the presacral fascia starting 5cm from the edge of the wound and pass to the other side 5cm from the edge of the wound including presacral fascia, subcutaneous tissue and the skin. Then pass 2cm from the edge of the wound and pass through the three layers to the other side in double u-shaped sutures. Multiple sutures are used according to the length of the wound. Sutures were approximated together without tension (Fig. 4-11).

   Group B:Rhomboid flap technique: involve closure of the defect after excision of all sinuses with Rhomboid flap of skin and subcutaneous tissue.

   Group C: Karydakis flap technique: the long axis of the ellipse is parallel to the midline and 2cm from it.undercutting incision is made along the whole length 1cm below the skin surface then unrolling the flap over the midline.

   Group D: Open procedure involved a wide excision of the pilonidal sinus tract and healing by secondary intention.

   2.2. Postoperative follow-up Postoperative management included pressure dressings, low residual diet until the fifth postoperative day, inspection of dressings in every other day, and suture removal on the 21th postoperative day. Instructions on discharge included avoidance of prolonged sitting and riding a bicycle until 8 weeks postoperatively to prevent wound disruption, improving local hygiene and regular removal of hairs by depilatory creams.

   Before discharge from hospital, patients are asked to return to the clinic on postoperative Day 3, Day 7, and Day 10. The skin sutures were removed on the 21th postoperative day. The long-term follow-up (1st month, 3rd month, 6th month, and 12th month) was performed via outpatient interview or by telephone interview.

   Successful treatment was the healing of the wound by subcutaneous scar formation and epithelization of the wound at 8-12 weeks. If skin and subcutaneous tissue reopened with discharge, it is reported as wound dehiscence. The wound that seemed to have healed within the first 8 weeks but recurred later on during the study period (either re-opening of a primarily healed pit or emerging of a new one) was documented as recurrence. A visual analogue scale (VAS) score was used to assess pain.
3. Statistical analysis:

Qualitative data were expressed as absolute frequencies (number) & relative frequencies (percentage). Categorical data were compared using Chi-square test. All tests were two sided. p-value < 0.05 was considered statistically significant. All data were collected, tabulated and statistically analyzed using SPSS 20.0 for windows (SPSS Inc., Chicago, IL, USA).

. 4. Discussion There is still no consensus about treatment of pilonidal sinus disease. Ideally, therapy should be associated with short hospital stay, less painful postoperative time, rapidly healing and return to work, less painful dressing of wound, short term wound care and a low recurrence rate. No techniques fulfill all of these criteria. We compared our results with other studies to estimate the reliability of our data.

Pilonidal sinus is more common in male [8]. In our study, male predominate than female (out of the total 160 patients 85% were males and 15% were females). Men are more affected thanks to their natural hirsutism.Most patients were young with the mean age in Group-A being 24.43 (SD ±6.08) and the mean age in Group-B was 27.40 (SD ± 5.90), Group C was 25.4 ± 5.3, Group D was 28.2±4.2. . Comparable results were shown in other similar studies [17].

Acute pilonidal abscess should be treated by incision and drainage. In the present study the patients presenting with an acute abscess in the sacrococcygeal region in 12 cases that were initially treated with incision and drainage then postoperatively they were treated by third generation cephalosporin and metronidazole for 10 days. Patients were scheduled for our technique after 15-30 days.

In a prospective randomized study performed on 50 patients and divided into two equal groups: drained and non-drained. Fluid collections were encountered in two patients (8%) of the drained group compared with eight patients (32%) in the no drained group with the difference being statistically significant [9].In our study, absence of wound collection, Seroma and hematoma in Group A and Group D are due to wide drainage by our special sutures technique and the use of third generation cephalosporin antibiotics, choosing non-infected pilonidal disease in most of cases.

A controlled study showed that wound problems, length of hospital stay, morbidity, and recurrence rates did not increase in the absence of postoperative draining of the cavity. Another study also demonstrated that drain placement after rhomboid excision and Limberg flap technique might negatively affect the postoperative complication rate, although the mean operation time was significantly longer in the non-drained group [10].In our study, we did not use drain in group A and the results showed decreased hospital stay, no Seroma nor hematoma , very low recurrence rate (2.5%) and infection occurred in one patient(2.5%).

In group A: most patients stopped analgesic drug on postoperative 3 days. Our patients started to sit on chair without pain on postoperative 10 days .It may result from low tension in the wound.

Primary closure technique's operation time is short but has significant postoperative morbidity as wound infection rate is 12-32.7%, dehiscence rate is 10- 50% and recurrence rate is 5-12% [11]. In this study, Group A showed infection in one patient(2.5%) and the recurrence rate was low (2.5%).

Incision and curettage, unroofing, curettage and excision with marsupialization procedures are common used surgical techniques. But these procedures had painful postoperative time, delayed healing and return to work, painful dressing of wound and long term wound care. But they have a low recurrence rate [12]. In this study, postoperative pain was low on pain scale, rapid wound healing, rapid return to work, and painless dressings and in addition, low recurrence rate (1%) When the midline lateralized or flattened, recurrences are less likely to occur [10].In our study there is partial flattening of the intergluteal cleft, and so the recurrence rate was low (2.5%).

Hospital stay varied from 2 to 5 days [13]. Using wide-excision techniques and median time off work was reported from 19 up to 38 days [14]. Other studies reported a mean length of hospital stay 2-4 days [9]. In the present study the length of hospital stay was 1 day in most cases of Group A and Group C.

The incidence of wound infection was ranged from 0% to 12% [15]. In our study, Group A showed Wound infection in one patient and Seroma did not occur in any patients.

Gupta [16] reported recurrence rates of 13% using wide-excision techniques, while other studies achieved 5% in larger trials [17]. A recurrence rate of 3-10% is described for excision with marsupialization of the wound [18]. Reconstructive flaps according to Limberg's technique come with a recurrence rate of 0-6% [13] in prospective randomized studies.

In classic Limberg flap technique recurrence rate is 1.26-5.3% [19]. In our study, Follow up time is 12 months and recurrence rate was in one case only (2.5%). Some studies have shown that, in addition to a good surgical technique, elimination of preventable risk factors such as hygiene at the intergluteal sulcus is important to prevent recurrence [20] [21].Therefore, patients in this study were advised regarding the importance of local hygiene.

Primary closure of the wound after excision of the pilonidal sinus is associated with a high recurrence rate. In the literature, the recurrence rate after primary closure has ranged from 4% to 25% [21].

A common complaint after flap surgery was hypoesthesia on the flap, in our study hypothesia occurred in 59 cases (37%).

Considering the problems of our study, there are two issues that have to be respected when interpreting our results: First, the recurrence rate of this study might be higher than demonstrated in the result due to shorter of follow up period and missing patients in the follow up period. Second, the wound healing time might have been shorter than it is reported in this study. The wound healing time was assessed by the patients themselves and was not determined by a physician. The wound healing time might more reflect the disappearance of any discomfort at the intergluteal fold than the complete closure of the skin after surgery.

ELIGIBILITY:
Inclusion Criteria:primary

* PSD in intergluteal region
* between 18-35 years.
* Also those fulfilling the diagnostic criteria of Chronic discharging sinus/sinuses in natal cleft with or without surrounding tissue inflammation and with associated pain and bleeding on clinical evaluation

Exclusion Criteria:

* recurrent pilonidal sinus,
* patients who were terminally ill, had Uncontrolled diabetics, were Immunocompromised and immunosuppressed patients,
* had acute pilonidal abscess.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
operative time | intraoperative
  operative time for all 4 groups are measured
infection postoperative | 2 weeks
  follow up the wound in early postoperative period

SECONDARY OUTCOMES:
postoperative recurrence | 1 year
  follow up the patient for 1 year to detect postoperative recurrence

IPD SHARING:
Plan to Share IPD: No
private data not for sharing